CLINICAL TRIAL: NCT03664739
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2 Arm, Parallel Group Study Comparing the Safety and Efficacy of IDP-120 Gel and IDP-120 Vehicle Gel in the Treatment of Acne Vulgaris
Brief Title: Study Comparing the Safety and Efficacy of IDP-120 Gel and IDP-120 Vehicle Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-120A-301
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2 Arm, Parallel Group Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As a double-blinded study, the investigators, the site staff, the sponsor, and the clinical monitors will not be aware of the treatment assigned to the individual study subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDP-120 Gel (Experimental): IDP-120 Gel, once-daily application
  Interventions: Drug: IDP-120 Gel
- IDP-120 Vehicle Gel (Placebo Comparator): IDP-120 Vehicle Gel, once-daily application
  Interventions: Drug: IDp-120 Vehicle Gel

INTERVENTIONS:
Drug: IDP-120 Gel — IDP-120 Gel, once-daily application
  Arms: IDP-120 Gel
Drug: IDp-120 Vehicle Gel — IDP-120 Vehicle Gel, once-daily application
  Arms: IDP-120 Vehicle Gel

SUMMARY:
study designed to assess the safety, tolerability, and efficacy of IDP-120 Gel and IDP-120 Vehicle Gel

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, tolerability, and efficacy of IDP-120 Gel and IDP-120 Vehicle Gel at Weeks 2, 4, 8, and 12. To be eligible for the study subjects must be at least 9 years of age and have a clinical diagnosis of moderate to severe acne

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 9 years of age and older;
2. Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit);
3. Subject must have a score of 3 (moderate) or 4 (severe) on the Evaluator's Global Severity Score (EGSS) assessment at the baseline visit;
4. Subjects with facial acne inflammatory lesion (papules, pustules, and nodules) count no less than 20 but no more than 50;
5. Subjects with facial acne non-inflammatory lesion (open and closed comedones) count no less than 25 but no more than 100;
6. Subjects with two or fewer facial nodules

Exclusion Criteria:

1. Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study;
2. Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram-negative folliculitis, dermatitis, eczema;
3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive;
4. Subjects with a facial beard or mustache that could interfere with the study assessments;
5. Subjects with more than two (2) facial nodules;
6. Evidence or history of cosmetic-related acne

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Companies
Locations (30):
- United States (25):
  - Valeant Site 123, Mobile, Alabama
  - Valeant Site 121, Hot Springs, Arkansas
  - Valeant Site 120, Beverly Hills, California
  - Valeant Site 117, Encinitas, California
  - Valeant Site 107, Fremont, California
  - Valeant Site 104, San Diego, California
  - Valeant Site 128, Denver, Colorado
  - Valeant Site 115, Wheat Ridge, Colorado
  - Valeant Site 113, Clearwater, Florida
  - Valeant Site 122, North Miami Beach, Florida
  - Valeant Site 103, West Palm Beach, Florida
  - Valeant Site 101, Oakbrook Terrace, Illinois
  - Valeant Site 124, Evansville, Indiana
  - Valeant Site 111, Louisville, Kentucky
  - Valeant Site 118, Largo, Maryland
  - Valeant Site 129, Needham, Massachusetts
  - Valeant Site 119, Detroit, Michigan
  - Valeant Site 126, New York, New York
  - Valeant Site 108, High Point, North Carolina
  - Valeant Site 106, Oklahoma City, Oklahoma
  - Valeant Site 109, Austin, Texas
  - Valeant Site 130, Pflugerville, Texas
  - Valeant Site 105, San Antonio, Texas
  - Valeant Site 110, Norfolk, Virginia
  - Valeant Site 116, Walla Walla, Washington
- Canada (5):
  - Valeant Site 112, Markham, Ontario
  - Valeant Site 102, Waterloo, Ontario
  - Valeant Site 114, Waterloo, Ontario
  - Valeant Site 125, Waterloo, Ontario
  - Valeant Site 127, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- IDP-120 Gel: IDP-120 Gel, once daily application
- IDP-120 Vehicle Gel: IDP-120 Vehicle Gel, once daily application
Period: Overall Study
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Started | 306 | 302
Completed | 256 | 270
Not Completed | 50 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel | Total
Number analyzed (Participants) | 306 | 300 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (7.6) | 20.5 (7.12) | 20.6 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 194 | 391
  Male | 109 | 106 | 215
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 16 | 15 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 75 | 65 | 140
  White | 197 | 202 | 399
  More than one race | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Lesion Counts at Week 12
Description: For noninflammatory facial lesions, open comedones (blackheads) and closed comedones (whiteheads) were recorded as a single count. For inflammatory facial lesions, papules (solid, elevated lesion less than 5 mm) and pustules (elevated lesion containing pus less than 5 mm) were recorded as a single count, while nodular lesions (palpable subcutaneous lesion greater than 5 mm) were counted and recorded separately.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: lesion counts
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 306 | 300
lesion counts
  Inflammatory lesions | -18.5 (10.79) | -13.3 (9.68)
  Non-inflammatory lesions | -26.3 (15.52) | -18.7 (14.28)

2. Primary Outcome: Percentage of Subjects Who Had at Least a 2-grade Reduction From Baseline at Week 12 in the Evaluator's Global Severity Score (EGSS) and Had an EGSS at Week 12 That Equated to "Clear" or "Almost Clear"
Description: Evaluator's Global Severity Score (EGSS) was determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations were scored on a scale of 0-4, with 0 being clear and 4 being severe.
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 306 | 300
percentage of participants | 41.7 | 20.4

3. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 12
Description: as for outcome 1
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 306 | 300
percentage change
  Non-inflammatory lesion count | -65.87 (37.467) | -47.54 (33.322)
  Inflammatory lesion count | -66.55 (35.017) | -48.64 (31.910)

4. Secondary Outcome: Percentage of Subjects Who Had at Least a 2-grade Reduction From Baseline at Week 12 in the Evaluator's Global Severity Score (EGSS)
Description: as for outcome 2
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 306 | 300
percentage of participants | 45.1 | 22.3

5. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 8
Description: as for outcome 1
Time Frame: Baseline to Week 8
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 306 | 300
percentage change
  Non-inflammatory lesion count | -56.06 (34.293) | -39.50 (33.217)
  Inflammatory lesion count | -60.07 (31.620) | -41.76 (30.710)

6. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 306 | 300
percentage change
  Non-inflammatory lesion count | -42.78 (32.109) | -30.73 (31.027)
  Inflammatory lesion count | -47.69 (32.010) | -35.23 (29.951)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: One subject was excluded from the safety population in the IDP-120 Gel group, due to not applying any study medication.
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/305 | 0/300
Serious Adverse Events (participants affected / at risk) | 1/305 | 0/300
Other Adverse Events (participants affected / at risk) | 27/305 | 3/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-120 Gel (N=305) | IDP-120 Vehicle Gel (N=300)
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-120 Gel (N=305) | IDP-120 Vehicle Gel (N=300)
Application site pain (General disorders) | 27 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT03664739/Prot_SAP_000.pdf